CLINICAL TRIAL: NCT01603966
Title: Low Dose Aspirin Study With the AggreGuide
Brief Title: Low Dose Aspirin Studied With the AggreGuide
Status: Completed | Type: Observational
Sponsor: Edward R. Teitel, M.D. (Industry)
Responsible Party: Sponsor-Investigator, Edward R. Teitel, M.D., CEO, Aggredyne, Inc.
Organization: Aggredyne, Inc. (Industry)
Other Study IDs: Val-030
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Platelet Aggregation
Keywords: platelet; aggregation; aspirin; inhibition; reactivity
MeSH Terms: conditions — Inhibition, Psychological

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: None Retained — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to determine whether the AggreGuide platelet aggregometer can discern the effect of low dose aspirin on subjects platelet aggregation using arachidonic acid as the agonist.

ELIGIBILITY:
Inclusion Criteria:

* adults

Exclusion Criteria:

* aspirin contraindications
* anticoagulants
* aspirin past week

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward R. Teitel, MD, Principal Investigator — Aggredyne, Inc.
Locations (1):
- Aggredyne, Inc., Houston, Texas, United States